CLINICAL TRIAL: NCT03691987
Title: Fecal Microbiota Transplantation in Chronic Fatigue Syndrome - an RCT
Brief Title: The Comeback Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: The Research Council of Norway (Other); Quadram Institute Bioscience (Other); Umeå University (Other); Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018/180
Record Dates: First submitted 2018-09-10; First posted 2018-10-02 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Chronic Fatigue Syndrome; Myalgic Encephalomyelitis
Keywords: fecal transplantation; bacterio therapy; fatigue; fecal microbiota transplantation
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preprocessed thawed donor FMT (Experimental): The active transplants are processed in a 2-3 weeks period before treatment of the first participant. Fifty to eighty grams of freshly delivered feces from donors is mixed with 100 mL isotonic saline and 25 mL 85% glycerol, homogenized and poured through a 0.5 mm mesh steel strainer, and transferred to 60 ml luerlock syringes and stored at -40°C.
  Frozen transplants are slowly thawed 2 hours prior to administration by transferring the FMT-syringes to a waterbath (+30°C). The transplant is then mixed with 125 mL 12°C isotonic saline in an enema bag prior to installation.
  Interventions: Biological: Preprocessed thawed donor FMT
- Preprocessed thawed autologous FMT (Placebo Comparator): The placebo transplant from each participant is prepared during the inclusion process four to six weeks before intervention and stored at -40°C. Fifty to eighty grams of freshly delivered feces from participants is mixed with 100 mL isotonic saline and 25 mL 85% glycerol is homogenized and poured through a 0.5 mm mesh steel strainer, and transferred to 60ml Luerlock syringes.
  Frozen transplants are slowly thawed 2 hours prior to administration by transferring the Luerlock syringes to a waterbath (+30°C). The transplant is then mixed with 125 mL 12°C isotonic saline in the enema bag prior to installation.
  Interventions: Biological: Preprocessed thawed autologous FMT

INTERVENTIONS:
Biological: Preprocessed thawed donor FMT — Delivered as an enema using the same equipment and technique as X-ray of the colon
  Arms: Preprocessed thawed donor FMT
Biological: Preprocessed thawed autologous FMT — Delivered as an enema using the same equipment and technique as X-ray of the colon
  Arms: Preprocessed thawed autologous FMT

SUMMARY:
This is a single-center stratified (on gender and donor), block randomized, placebo-controlled, parallel group trial with 12-months follow-up of 80 chronic fatigue syndrome/encephalomyelitis (CFS/ME) participants. Participants will be randomized to treatment by preprocessed thawed donor fecal microbiota transplant or preprocessed thawed autologous fecal microbiota transplant. Primary endpoint is the efficacy of FMT at three months by the Fatigue Severity Scale. The investigators will use patient reported outcomes for primary and secondary outcome measures.

Previous studies suggest that a dysbiosis of the gut microbiota may be a key feature in CFS/ME. We hypothesize that

A: CFS/ME is caused by a dysbiosis in the gut flora causing barrier leakage of bacterial products, a low grade systemic immune activation and disturbances in the host energy metabolism.

B: Recovery of a normal gut flora by fecal microbiota transplantation (FMT) alleviates symptoms and may even induce remission of CFS/ME.

This project aims to determine if there is a true cause and effect relationship between a dysbiotic gut flora and CFS/ME by testing if treatment of the observed dysbiosis by FMT also can resolve CFS/ME symptoms. In this process, collection of blood, fecal, and urine samples before and after FMT will open the possibility to explore the relationship between the gut flora, immune response, host energy metabolism and CFS/ME using technologies of microbiomics, metabolomics and immunological characterizations for a better understanding of the pathobiology of CFS/ME.

DETAILED DESCRIPTION:
CFS/ME participants:

General practitioners recruit participants from the local area, by posters at the doctors' offices. In addition the study has a facebook site, named "the COMEBACK study", where interested CFS/ME subjects can submit their interest to be assessed for participation. After a telephone screening of potential participants by the International Consensus Criteria for CFS/ME and CFS/ME severity rating, eligible subjects will be referred to department of physical medicine and rehabilitation UNN Harstad (FYSMED) and re-assessed. During this screening process the investigators will keep a track record of screening failures noting reason for failure. Participants will have a physical exam and necessary workup including blood, fecal and urine tests to exclude differential diagnosis according to the Norwegian National Guidelines for Assessment of CFS/ME. Participants receive information about the study and give their written consent. Subjects earlier diagnosed with CFS/ME at FYSMED will undertake the same re-assessment.

During the work up, participants will do the Fatigue Severity Scale, Hospital Anxiety and Depression scale, SF 36, Modified DePaul Questionnaire, the Rome IV criteria for irritable bowel syndrome, and the "Repeatable Battery for the Assessment of Neuropsychological Status" test (RBANS). Heart rate variability is implemented as an additional measure when approximately 40 out of 80 participants are assigned treatment.

Donors are recruited informally from the local high schools. Donors are included and screened according to the European Consensus Guidelines from 2017. The full screening will be undertaken before the first feces donation and every 4th week. The inclusion and screening will be performed at the department of physical medicine and rehabilitation UNN Harstad. The investigators will keep a track record of screening failures noting reason for failure.

Participants receive FMT at the gastroenterology outpatient clinic at University Hospital of North Norway Harstad, Norway. No antibiotics are given prior to the intervention. The participants must do a bowel lavage using Sodiumpicosulphate/Magnesiumcitrate (Picoprep, Ferring) before intervention. The treatment will be administered by enema. Active treatment will be pre-processed frozen donor feces. Placebo will be the participant's own feces processed and frozen during the study inclusion. After the intervention, the participants have no restrictions on activity level and are asked to keep an unchanged diet without introduction of any new food supplements or probiotics in the follow up period. To keep track of change in diet investigators ask participants to do a food frequency questionnaire before the FMT and at 3 and 12 months after the intervention. Use of antibiotics, food supplement and use of medications will also be recorded.

The treatment will take place in blocks of four consecutive participants per day. A data engineer at the Department of Clinical Research at the University Hospital of North Norway, Tromsø (UNN,Tromsø) creates the allocation sequence using the REDCap software. The treatment is randomized on donor and placebo in fixed blocks of 4 with 2 active (1 donor A and 1 donor B) and 2 placebo. Block allocation will be stratified on gender.

A stratification on donor and gender will be performed by assigning full blocks of male and female participants. In the two active slots in each block of four, one active slot will be used for donor A and one for donor B. The stratification of gender reflects the higher incidence of CFS/ME in women. Donor fecal microbiota transplants stored for more than two years will be disposed and replaced with transplants from a new donor. If this happens, donor fecal microbiota transplants from the new donor will be assigned in remaining slots from the donor with the expired transplants.

Allocation is done in solitude in a closed room with no transparency, only containing a freezer with the active transplants (tagged by donor batch ID) and the placebo transplants (tagged by screening number). Before allocation of treatment, an investigator places the FMT-placebos on a table in the room. The allocator can then enter the room as the researcher placing all the placebos leaves the room. The allocator will access the randomization sequence when entering participants screening number on the REDCap software using a computer in the same room. The allocator will be the only person involved in the study that can access the randomization program at the REDCap software. If a screening number is randomized to active treatment, the allocator removes the tag from the placebo and places it on a donor FMT treatment instead. All unused placebo transplants will be disposed immediately. When finished, the allocator places the allocated treatment in a box in a designated freezer. The allocator will build a key file matching the active treatment to the donor batch id by updating a key file on paper and store it in a safe not accessible to any others. In addition the allocator will write the corresponding patient screeningnumber on tags from the used donor batch and keep them as backup in the same safe. This will allow for tracking of each individual donor batch to a corresponding participant at the end of trial when all follow up is complete.

ELIGIBILITY:
FMT PARTICIPANTS

Inclusion Criteria:

* International Consensus Criteria for CFS/ME
* 18-65 years
* Mild-severe CFS/ME
* Fatigue Severity Scale score of 5,0-7,0
* Symptom duration for 2-15 years

Exclusion Criteria:

* Kidney failure
* Congestive heart failure
* Immuno-deficiency or use of immune-suppresive drugs
* Other disease that may explain ME/CFS symptoms discovered during diagnostic work up
* Use of antibiotics the last three months,
* Use of low dose naltrexone or Isoprinosin
* Pregnancy or breastfeeding
* Serious endogenous depression
* Chronic infectious disease (HIV, hepatitis B or C etc.)
* Introduction of new food supplements, change in diet or introduction of new medications the last three months
* Assessed not be able to follow the instructions for data and sample collection
* Very severe ME/CFS (WHO class IV)
* Symptom duration of less than 24 months or more than 15 years
* History of abdominal surgery, with the exception of appendectomy, cholecystectomy, caesarean section and hysterectomy
* Previous treatment with FMT

FMT DONORS

Inclusion criteria:

* Healthy
* Age 16-30 years
* Type 3 or 4 stool by the Bristol Stool Scale

Exclusion criteria:

* Use of peroral antibiotics past 3 months
* Use of topical antibiotics past 2 months
* Tattoo or piercing past 6 months
* Former imprisonment
* History of: -chronic diarrhea
* constipation
* inflammatory bowel disease
* colorectal polyps
* colorectal cancer
* immuno-suppression
* Obesity
* Metabolic syndrome
* Atopic skin disease
* CFS/ME
* Psychiatric disorders
* Other serious autoimmune disease
* Close relatives with serious autoimmune disease
* High risk sexual behavior
* Bowel movements that does not correspond to a Bristol Stool Scale type 3 or 4
* Journeys abroad the last six months to countries high in antibiotic resistance
* Use of food supplements, pre-, -pro, -or symbiotics past one month
* Dysbiosis grade 3 or more by the GA dysbiosis test

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion with treatment success in FSS score in donor versus placebo FMT group. Treatment success is defined as an improvement of more than 1.2 points on the Fatigue Severity Scale (FSS) | Three months after treatment
  Fatigue Severity Scale (FSS) is a self-reported, 9-item fatigue scale. Participants rate all 9 items on a 7-point Likert scale (1-2-3-4-5-6-7) depending on how appropriate they felt the statement applied to them over the preceding week. The total score is calculated by adding up the answer from each item and divide by 9. Lower scores indicate better outcomes. Maximum score is 7.
  In an intention to treat analysis we will categorize participants as responders/non-responders, defining responders as decrease of more than 1,2 to the total baseline score in the FSS at 3 months post FMT by Chi Square. Baseline score will be the average of the two scores from the screening period. Missing values will be regarded as non responders

SECONDARY OUTCOMES:
Change in donor versus placebo FMT group in fatigue by the Fatigue Severity Scale score | Change in Fatigue severity scale by repeated measures from baseline and until 1, 3, 6, 9 and 12 months after treatment
Change in donor versus placebo FMT group in quality of life by the SF36 score | Change in SF36 score by repeated measures from baseline and until 3 and 12 months after treamtent
  The SF-36 consists of eight scaled scores (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health), which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Change in donor versus placebo FMT group in neurocognitive function by the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) score from baseline and until 3 months after treatment. | Change from baseline and until three months after treatment
  RBANS is a neuropsychological assessment that consists of ten subtests which give scores to five domains: Immediate memory, visuospatial/constructional ability, language, attention and delayed memory.
Change in donor versus placebo FMT group in anxiety and depression by the Hospital Anxiety Depression Scale (HADS) score | Change in HADS score by repeated measures from baseline and until 3 and 12 months after treatment
  HADS is an instrument with 14-items for detection of depression and anxiety in hospitalized patients. Scores range from 1-21 interpreted as: normal (0-7), mild (8-10), moderate (11-14), severe (15-21). Subscales for anxiety (HADS-A) and depression (HADS-D) is also defined. We will explore the FMT effects on HADS by an independent sample T-test (or, if necessary, non-parametric Mann-Whitney) comparing change in global score. We will apply last value forward for missing values.
Change in donor versus placebo FMT group in gastrointestinal related complaints by the sum score of selected items in the DePaul Questionnaire (DPQ) (29, 30, 46 and 47) | Change in DPQ score by repeated measures from baseline and until 6 and 12 months after treatment
  The DPQ assesses key symptoms of ME/CFS such as fatigue, gastrointestinal complaints, post-exertional malaise, sleep, pain, neurological/cognitive impairments and autonomic, neuroendocrine and immune symptoms. At each item, participants have to rate the frequency and severity of the symptom on a scale from 0 to 4. We wil use the sum score from the questions that assess gastrointestinal complaints in the DPQ in this endpoint. This endpoint was implemented after 19 out of 80 participants had completed the three months follow up
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Baseline to end of follow up at 12 months after FMT
  Participants will be screened for adverse events from the time of informed consent through the end of the trial. In case of an identified adverse event, this will be recorded and described in the CRF
Change in HRV in donor FMT vs placebo FMT group derived from the R-R intervals in continuous ECG recordings. The primary vagal function outcome will be differences in changes from pre-post treatment between groups in High Frequency HRV (HF-HRV; in ms2 | 3 months after treatment
  Firstbeat Bodyguard will record R-R interval and the Firstbeat life style assessment software will analyze the R-R interval recording and provide the outcome measure
Change in HRV in donor FMT vs placebo FMT group derived from the R-R intervals in the resting continuous ECG recordings. The secondary vagal function outcome will be differences in changes from pre-post treatment between groups in RMSSD (RMSSD; in ms2) | 3 months after treatment
Difference in mean baseline HRV (HF-HRV and RMSSD) between responders vs non-responders to donor FMT. | 3 months after treatment
  As defined by the primary endpoint in the clinical study, a responder will be defined as an improvement of more than 1.2 points on the Fatigue Severity Scale (FSS) from baseline and until 3 months after treatment. To determine HRV in each group we will use High Frequency Power analysis denominating HRV in ms2.

OTHER OUTCOMES:
Engraftment of donor microbiota | 3 months after FMT
  Comparison between baseline profile, post FMT and donor profile will show if engraftment of donor mikrobiota parallels clinical response to active FMT. To assess fecal gut microbiota composition, morning stool samples will be obtained at baseline and three and twelve months after FMT. Participants will collect their first morning bowel movement in a 120ml container for storing in their home freezer (-20C). Two-four weeks after, samples will be collected from participants home and stored on dry ice during transport until freezing at -80°C at the University Hospital of North Norway Harstad. Fecal analysis will be done by NextSeq500 allowing for enhanced metagenomics (prokaryote and viral) sequencing.
Engraftment of donor microbiota | 12 months after FMT
  Comparison between baseline profile, post FMT and donor profile will show if engraftment of donor microbiota parallels clinical response to active FMT. To assess fecal gut microbiota composition, morning stool samples will be obtained at baseline and three and twelve months after FMT. Participants will collect their first morning bowel movement in a 120ml container for storing in their home freezer (-20C). Two-four weeks after, samples will be collected from participants home and stored on dry ice during transport until freezing at -80°C at the University Hospital of North Norway Harstad. Fecal analysis will be done by NextSeq500 allowing for enhanced metagenomics (prokaryote and viral) sequencing.
Difference in metagenomic profile between responders and non responder to FMT | Baseline samples before FMT
  To assess fecal gut microbiota composition, morning stool samples will be obtained at baseline and three and twelve months after FMT. Participants will collect their first morning bowel movement in a 120ml container for storing in their home freezer (-20C). Two-four weeks after, samples will be collected from participants home and stored on dry ice during transport until freezing at -80°C at the University Hospital of North Norway Harstad. Fecal analysis will be done by NextSeq500 allowing for enhanced metagenomics (prokaryote and viral) sequencing.
Change in the nature of host immune and antibody response | Change from baseline to 3 months and difference between responders and non-responders to treatment at 3 months
  Analysis (multipex technology) of mediators in the innate and adaptive immune response
Change in the nature of host immune and antibody response | Change from baseline to 12 months and difference between responders and non-responders to treatment at 12 months
  Analysis (multipex technology) of mediators in the innate and adaptive immune response
Difference in the nature of host immune and antibody response between responders and non responders to FMT | Baseline samples before FMT
  Analysis (multipex technology) of mediators in the innate and adaptive immune response
Change in the metabolome in feces, blood and urine | Change from baseline to 3 months and difference between responders and non-responders to treatment at 3 months
  Analysis (mass spectrometry) on fecal extracts, urine and serum in order to assess the functional output of the microbiota
Change in biomarkers for breach in gut epithelium (sLPS-binding protein and sCD14) before and after transplantation | Change from baseline to 3 months and difference between responders and non-responders to treatment at 3 months
  Analysis (ELISA) of immunological markers associated with gut barrier leak (sCD14 and sLPS-BP)
Change in biomarkers for breach in gut epithelium (sLPS-binding protein and sCD14) before and after transplantation | Change from baseline to 12 months and difference between responders and non-responders to treatment at 12 months
  Analysis (ELISA) of immunological markers associated with gut barrier leak (sCD14 and sLPS-BP)
Difference in biomarkers for breach in gut epithelium (sLPS-binding protein and sCD14) in responders and non responders to FMT | Baseline samples before FMT
  Analysis (ELISA) of immunological markers associated with gut barrier leak (sCD14 and sLPS-BP)

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus Goll, MD. PhD., Principal Investigator — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Harstad, Harstad, Troms, Norway

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Available when findings from primary and secondary endpoints are published. Study protocol will be available upon request when we initiate the inclusion.
Access Criteria: Data access requests will be reviewed by study investigators. Requestors will be required to sign a Data Access Agreement

REFERENCES:
- [Derived] Skjevling L, Goll R, Hanssen HM, Johnsen PH. Faecal microbiota transplantation (FMT) in Norwegian outpatients with mild to severe myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS): protocol for a 12-month randomised double-blind placebo-controlled trial. BMJ Open. 2024 Jun 10;14(6):e073275. doi: 10.1136/bmjopen-2023-073275. PMID 38858151